CLINICAL TRIAL: NCT02236117
Title: The Effects of 10 Weeks of Aerobic Training on the Autonomic Modulation in Prepubertal Children: a Randomized Control Trial
Brief Title: Aerobic Training on the Autonomic Modulation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Carla Cristiane da Silva, The Effects of 10 weeks of aerobic training on the autonomic modulation in prepubertal children: a randomized control trial, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CONEP 5231
Record Dates: First submitted 2014-08-25; First posted 2014-09-10 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Healthy
Keywords: heart rate variability; children; progressive test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Aerobic Training (Experimental): The children included in the experimental group will make 10 weeks of aerobic training. The intensity of the race will be based on individual speed obtained in the last stage completed the progressive test, known as the maximal aerobic speed (MAV) in km/h. The running speed of the exercise protocol will be minimum 80% of the MAV in the protocol of continuous training. The intermittent progressive training is n * (10*15 s) to 100% MAV, and n from 2 to 6 series between the first and tenth week. The training protocol was adapted from previously described (Mandigout et al, 2002, Gamelin et al, 2009.). Acceptance of the exercise in a pediatric population has been previously observed by pilot study.
  Interventions: Other: Aerobic Training
- physical education classes (No Intervention)

INTERVENTIONS:
Other: Aerobic Training — Will be included 160 children, 80 in an experimental group and 80 in a control group of both genders. The experimental group will realize aerobic training during 10 weeks (3×40min week-1; intensity, >80% maximal aerobic velocity - MAV), while the control group will have involved with the physical education classes two times a week for 50 minutes each class. The aerobic protocol will be composed by 2 sessions of intermittent running and 1 session by continuous.
  Arms: Intervention: Aerobic Training

SUMMARY:
The heart rate variability is a tool used to asses non-invasive cardiac autonomic. In fact, many studies have been disseminated of heart rate variability in adults, however few results in a literature this parameters in pediatric population, mainly with children submitted the physical training. Thus, this Project aims to verify the effects of aerobic training, with 10 weeks, in prepubertal on the performance and heart rate variability in rest.

DETAILED DESCRIPTION:
The randomized control trial in accordance with Consort - Statement (Moher et al., 2012) will be done. Will be included 160 children, 80 in an experimental group and 80 children with no intervention, of both genders.

ELIGIBILITY:
Inclusion Criteria:

* Children be with body weight and height between the 10th and 90th percentiles, according to criteria adopted by the Centers for Disease Control and Prevention (CDC, 2002).
* To characterize the infant state, all volunteers will conduct evaluation of secondary sexual characters by criteria of Tanner (Marshall and Tanner, 1970), through visual inspection by a single experienced paediatrician. Children must show the initial stage of pubertal development, for girls (1 breast) and boys (genital 1) to be included and characterized such prepubertal. Participants throughout the trial entering puberty will be excluded from the final analysis.
* The children will be healthy, without clinical or historical evidence of cardiovascular disease, hypertension, insulin-dependent diabetes mellitus or obesity, and were not taking any drugs.

Exclusion Criteria:

* The participants can be not linked to sports practices at least one year before the beginning the study, and can be involved only with the physical education classes two times a week for 50 minutes each class.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Rest Heart Rate Variability in short term | 10 weeks
  The cardiac autonomic modulation of the sinoatrial node will be estimated via heart rate variability (HRV) pre- after 5 weeks - post-10 weeks of training and after 8 weeks of finished the intervention (follow-up period). The duration of the RR interval recordings (RRinterval) will be obtained from each children using a portable heart rate monitor (Polar RS800) at a sampling rate of 1000 Hz. The recordings will be downloaded via commercial software and export for later analysis of time and frequency domain measures of HRV. The time domain indices examined will be: the mean RR interval, the root-mean-square difference of successive normal RR intervals (RMSSD), which reflects vagal modulation, and the standard deviation of all normal RR intervals (SDNN), which comprises both sympathetic and vagal cardiac modulations (Task Force, 1996).

CONTACTS AND LOCATIONS:
Overall Officials: Carla Silva, Doctor, Principal Investigator — Universidade Estadual de Londrina
Locations (1):
- Universidade Estadual de Londrina, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No